CLINICAL TRIAL: NCT06817993
Title: Development of a New Social Media fMRI Task to Better Investigate Bidirectional Links Between Social Media Use and Emotional Health in Youth
Brief Title: Teen Brain Online II: Understanding How Social Media Affects the Teen Brain
Acronym: TBO-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Silk, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY24100085; 1R21MH138955-01 (NIH)
Record Dates: First submitted 2024-12-20; First posted 2025-02-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: Depression; Adolescent; Teen; Social Media; Social Acceptance; Social Rejection; fMRI; Neuroimaging
MeSH Terms: conditions — Depression; Social Isolation

STUDY DESIGN:
Intervention Model Description: All participants will be similar (13-17 with at least mild depression symptoms) and will experience the same procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adolescents aged 13-17 with at least mild symptoms of depression (Experimental): Adolescents in Phase 2 will be screened for depressive symptoms using the MFQ-c. 20 teens will have MFQ-c scores within the mild range (MFQ = 12-25). The sample will be stratified, with 30 teens who will have moderate to severe depressive symptoms as assessed by the MFQ-C. (MFQ ≥25; N=30)
  Interventions: Behavioral: Rejection and Acceptance Feedback

INTERVENTIONS:
Behavioral: Rejection and Acceptance Feedback — Participants will be administered cues of peer acceptance and rejection from virtual peers during an fMRI task. In the CHAT-I task, they will be chosen or not chosen to discuss various topics with a virtual peer. In the TBO Task, they will receive a high or low number of likes relative to the other photos displayed of peers. They will also view comments on their posts from peers, which may have positive, negative, or neutral content.

SUMMARY:
There has been much interest in the potential role of social media (SM) use in driving a current mental health crisis among teens, with a dire need for evidence that goes beyond self-report. One important avenue is to understand the role of the brain in driving the effects of SM use on emotional health and vice versa. However, there is almost no research addressing these questions, largely due to a lack of tasks that can probe the neural correlates of modern SM use. The goal of this clinical trial is to develop and validate a new developmentally-appropriate and ecologically-valid functional magnetic resonance imaging (fMRI) and eyetracking task, the TeenBrainOnline (TBO) Task, that is more realistic and similar to modern SM platforms. Participants will be 50 teens (ages 13-17) with depressive symptoms who will complete the final version of TBO task during fMRI with eye-tracking, an older Chatroom Interact (CHAT-I) Task, daily surveys of SM use, and measures of depressive symptoms. Our goal is to show that the task works by:

* Demonstrating that it activates expected regions of the brain and visual attention biases toward feedback cues.
* Showing that brain and eyetracking (visual attention) activity on the task explain variability in depressive symptoms at baseline and three months later, and work better than similar indices from an older task.
* Showing that brain and eyetracking (visual attention) activity on the task are associated with real-world measures of social media use collected during daily surveys. Specifically, The investigators expect that teens whose brain and eyetracking activity suggests they are more sensitive to feedback on SM will report a social evaluation orientation toward social media use in daily life, such as engaging a lot in social comparison, worrying about missing out, and caring about getting a lot of likes and comments.

Participants will be asked to:

* complete a 10-15 minute screening call to determine eligibility for the study
* complete one 90 minute virtual study visit to complete questionnaires and prepare for the MRI visit (visit 1)
* submit 24 photos to our study specific social media site
* complete an (in person) MRI scan visit (~4 hours), which consists of 2 tasks where they will interact with peers (visit 2)
* complete ~5 minute smartphone surveys 3 times a day for 16 days, asking about their daily experiences online and emotional reactions.
* complete 2 online questionnaires asynchronously 3 months after their scan date

DETAILED DESCRIPTION:
There is no assignment to conditions. All participants will receive the same intervention, which is the completion of two experimental tasks that present participants with opportunities to receive feedback from peers. Phase 1 focuses on task development with 10 participants, where they will complete a screening call, a 60 virtual screening call with questionnaires and preparation for the fMRI tasks (TBO and CHAT) described below. They will then complete the Teen Brain Online (TBO) and Chatroom Interact (CHATI) tasks during fMRI/eye-tracking at the BRIDGE MRI Center in a counterbalanced order (with half of the participants randomly assigned to complete the CHAT task first, and the other half randomly assigned to complete the TBO task first), approximately one month following the screening visit. Phase 1 participants will not have EMA text message surveys or a 3 month follow up visit. During Phase 2 (~months 9-24), the final version of TBO will be tested in 50 youth with elevated depressive symptoms. Following a phone screen, youth will complete a virtual screening visit that includes questionnaires and preparation for the fMRI tasks. They will then complete the Teen Brain Online (TBO) and Chatroom Interact (CHATI) tasks during fMRI/eye-tracking at the BRIDGE MRI Center in a counterbalanced order, approximately one month following the screening visit, as well as measures of depressive symptoms at three months (Mood and Feelings Questionnaire (MFQ).

Before the MRI visit, youth are asked to submit 24 selfies, a profile picture, and a handle for a study specific social media site All participants will get a chance to view the site before their MRI scan to view and interact with posts, through likes and comments systems. During the TBO task within the scanner, the participants will be shown their own posts and the posts of other teens in the study alongside each other. They will also be shown the number of likes, comments, and views on each post. The investigators will assess their neural reactions to the posts, and also use eye tracking to see what they are paying attention to on screen. The Investigators will also assess the teen's reactions to 3 of their posts comment's sections. In the inter-block intervals, the investigators will also show them trials with 2 peer photos to control for the effect of seeing images of peers vs themselves. The placement of participant and peer photos are random (left vs right), and no photos will be repeated.

For the CHAT-I Task, participants will view photos and biographies for same-age youth and choose the top five that they would like to interact with from other research sites. They will have their own photo taken (via screenshot) and provide a biography for their own profile. They will be matched with two of the five available peers, and will interact with them in the scan. During the CHAT-I task in the scanner, the participant and peers take turns selecting who they would rather talk to about a series of topics (e.g., music, movies). The first block is a neutral condition in which a dot appears over the picture of one person, and the participant presses a button indicating on which side the dot appeared. The chat game then proceeds in three blocks, where the participant and the peers will take turns selecting who they would like to talk to.

Teen participants will also complete a 16-day EMA protocol (two school weeks, three weekends) using Web-DataExpress. This approach will allow us to obtain nuanced information about SM experiences beyond frequency/duration of use. Following our standard procedures, they will be randomly sampled within three blocks of time (morning, after school, evening) for a total of 48 surveys. Youth can "snooze" each prompt for up to one hour, and the after-school prompt allows youth to report SM use during the school day.

Certain information is withheld to protect the scientific integrity of the study design.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 13-17
* Depression screening scores on the MFQ-C in the mild (MFQ = 12-25; N = 20) or moderate-to-severe range (MFQ ≥25; N=30)
* Possess their own smartphone to complete web-based ecological momentary assessments (EMA) using WebDataExpress.
* use social media apps (e.g. Instagram, twitter, reddit, discord, YouTube, etc.) at least 3 times a week, on average, per teen report

Exclusion Criteria:

* Presence of a serious neurological or medical condition, by parent report
* Unable to read or speak English or cognitive impairment preventing ability to complete assessments.
* Hearing impairment preventing ability to hear and understand instructions conveyed via headphones in the MRI scanner
* Possible pregnancy, as determined by participant report
* Presence of probable substance use disorder, as determined by participant report
* Presence of MRI contraindications (e.g., dental braces, history of metallic foreign objects in body such as aneurysm clips or other devices or questionable history of metallic fragments, claustrophobia, or a weight of above 300 lbs)
* Taking medications that affect the central nervous system other than antidepressants (stable dose allowed due to high rates of use among teens with depressive symptoms) or stimulants if required 36 hours before the scan.
* Completion of Chatroom Interact Task or TBO Task in prior studies
* Screening positive on the Autism Spectrum Screening Questionnaire, or screening positive on the Youth Inventory-4/ for a potential psychotic disorder or substance use disorder.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Average Affective Salience Network Activation to Social Reward and Threat stimuli | During the MRI Scan/intervention (occurring once ~4 weeks into the study)
  The investigators will measure neural activity (as measured by fMRI response) in regions within the Affective Salience network (ASN) in response to social threat and reward in the TBO and CHAT-I tasks. Average activation will be compared in each region between experiences of social reward, social threat, and neutral experiences as well as baseline.

SECONDARY OUTCOMES:
Depressive Symptoms Score as Assessed by the MFQ-C | baseline (phone screen), immediately before the Intervention, 3 months
  Depressive symptoms are measured measured by the Mood and Feelings Questionnaire-child. (MFQ-c), at baseline at a screening call, concurrently at the time of scan visit, and at 3 months. Scores on this assessment are measured continuously and will be assessed for their correlation with other outcome measures.
Average Visual Fixation time to Social Reward and Threat stimuli | During the MRI Scan/intervention (occurring once~4 weeks into the study)
  The Investigators will measure eye-tracking fixations of over 50 ms to areas of interest (AOIs) in the TBO task, including the self-photo, other-photo, likes, views and comments numbers, and the comments themselves. Gaze duration will be computed for each AOI divided by the total length of the trial for each condition, then average gaze durations across all trials within each condition (reward, threat, neutral).
Reported Emotional Experiences of Threat and Reward during Daily Social Media Use | 3 times a day for 16 days
  Participants will be asked to select which SM apps they used since their last survey, and their reported passive/active behaviors, using validated items from Common Sense Media. They will then rate several aspects on a 0-100 slider. They will rate social comparison orientation using an item adapted from Nesi's Emotional Responses to SM Scale - Revised. Digital status seeking will be assessed using behaviors from Nesi's digital status seeking measure. Online FoMO will be assessed with items from the online adaptation of the FoMO scale. Affective responses to SM will be assessed by having youth nominate their most positive and negative experiences via SM since the last survey and rate their associated positive affect (PA; average of "happy," "joyful," "interested," "excited") and negative affect (NA; average of "worried," "stressed," "mad", "sad").

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Silk, Ph.D, Principal Investigator — University of Pittsburgh; Helmet T Karim, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the study, after deidentification, may be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Scientific data will be made accessible no later than 1 year after the grant end date. Any subject level data and associated analyzed data will be shared at time of publication. No end date.
Access Criteria: Deidentified data will be submitted to and made available on the National Institute of Mental Health Data Archive (NDA). To obtain data access, researchers will follow the established procedures within NDA, and the NDA Data Access Committee will determine the approvals for these requests. Access will be given for any legitimate scientific purpose, as determined by NDA Access Committee.